CLINICAL TRIAL: NCT04805866
Title: Tracking Neural Synergies During Gait Rehabilitation After Stroke
Brief Title: Tracking Neural Synergies After Stroke.
Status: Active, not recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigaor, Shirley Ryan AbilityLab
Other Study IDs: STU00214290
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Electromyography; Gait rehabilitation; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Age-matched controls: Healthy individuals ages 18-85
- Inpatients poststroke: Individuals post acute or subacute that that are inpatients at the Shirley Ryan AbilityLab ages 18-85

SUMMARY:
The purpose of this study is to identify neural muscle synergies of patients post-stroke and track them during an inpatient acute rehabilitation. To this end, the researchers will use an innovative approach based on the identification of large populations of motor units from recordings of surface high-density electromyography (HD-EMG).

DETAILED DESCRIPTION:
The researchers will focus on the identification of neural muscle synergies of leg and thigh muscles during postural and locomotor tasks in patients post stroke. To this end, the researchers will recruit 20 patients participating in inpatient rehabilitation at Shirley Ryan AbilityLab in the early subacute phase after stroke and 20 age-matched healthy controls. The researchers will ask them to perform postural tasks and walking trials at their preferential speed. All assessments will be performed by a licensed physiotherapist as per the standard of care once a week during three weeks of inpatient rehabilitation at the Shirley Ryan AbilityLab. During these tasks, the researchers will record HD-EMG signals from four muscle groups (Quadriceps, Hamstrings, Triceps Surae, Tibialis anterior).

ELIGIBILITY:
Healthy participants:

Inclusion Criteria:

* Age 18-85 years old
* Ambulatory with or without an assistive device
* Ability to stand unassisted for at least 15 min
* Informed consent provided by participant
* English speaking

Exclusion Criteria:

* Inability to communicate with researchers
* Lower extremity joint pain, contractures
* Major sensory deficits, or cardiovascular or respiratory symptoms contraindicative of walking
* History or evidence of orthopedic, muscular, or physical disability
* Taking current medications that may affect balance
* History or evidence of vestibular, auditory, or proprioceptive impairment
* History or indication of orthostatic hypotension
* History of any neurological disease
* Open wounds on surfaces in contact with HD-EMG electrodes
* Concurrent participation in other lower limb research studies that according to the PI is likely to affect study outcome or confound results
* Pregnancy

Patients:

Inclusion Criteria:

* Age 18-85 years old
* Unilateral, supratentorial ischemic or hemorrhagic stroke within the past six months
* Medical clearance from primary medical team (signed Medical Clearance form)
* Unassisted sitting balance at edge of mat or hospital bed ≥ 30 seconds
* Baseline Visible muscle contraction in hip flexors, knee extensors, and ankle dorsiflexors ( ≥1 MMT) or manual resistance against one muscle group (>3 MMT)
* Adequate cognitive function as determined by the NIH scale: score ≤1 on question 1b and score =0 on question 1c
* Informed consent provided by participant or POA
* English speaking

Exclusion Criteria:

* Severe aphasia limiting ability to express needs or discomfort verbally or nonverbally
* Severe behavioral neglect
* History of prior stroke
* Concurrent neurologic condition (i.e PD, TBI, MS, etc.)
* History of peripheral nerve injury
* Joint contracture or significant spasticity in the lower limbs (Modified Ashworth Scale ≥3)
* Severe knee, hip, or ankle osteoarthritis
* Severe osteoporosis as indicated by physician medical clearance
* Open wounds on surfaces in contact with HD-EMG electrodes
* Unstable spine or unhealed fractures
* Weight bearing precautions
* Unresolved deep vein thrombosis (DVT)
* Concurrent participation in other lower limb research studies that according to the PI is likely to affect study outcome or confound results
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals poststroke that are inpatients at Shirley Ryan AbilityLab and Healthy individuals as age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neural Synergies | Baseline and Once weekly, through completion of study up to 4 weeks
  The neural synergies are group of muscles that receive a common input from the brain. The researchers will assess the common input as the level of correlated activity between muscles. The researchers will compare this level of correlated activity between legs and groups, and how this changes over the course of the study

SECONDARY OUTCOMES:
10 Meter Walk Test | Baseline and Once weekly, through completion of study up to 4 weeks
  The 10 Meter Walk Test is a common clinical measure of gait speed. Participants will be directed to walk at their comfortable, self-selected speed. Participants will be positioned at the start line and instructed to walk the entire 10 meter distance while the therapist times the middle six meters. The distance before and after the timed course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.46 sec). The test will be performed two times at self-selected speed with adequate rest in between. The average of the two times should be recorded. The test will then be repeated with the participants directed to walk at their fast but safe speed. Appropriate assistive devices, bracing, and the minimal amount of physical assistance from the physical therapist will be applied.
6 Minute Walk Test | Baseline and Once weekly, through completion of study up to 4 weeks
  The 6 Minute Walk Test measures the distance a participant can walk indoors on a flat, hard surface in a period of six minutes. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test is self-paced. Participants are allowed to stop and rest during the test; however, the timer does not stop. If a participant is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. Appropriate assistive devices, bracing, and the minimal amount of physical assistance from the physical therapist will be applied.
Berg Balance Scale | Baseline and Once weekly, through completion of study up to 4 weeks
  The Berg Balance Scale is a 14-item test, scored on a five point ordinal scale. It measures functional balance in a clinical setting and includes static and dynamic tasks (such as sitting, standing, transitioning from sitting to standing, standing on one foot, retrieving an object from the floor), during which participants must maintain their balance.
Quality Indicators | Baseline and Once weekly, through completion of study up to 4 weeks
  This is a standardized, evidence-based measure of health care quality used to track clinical performance and outcomes in post-acute care. Items are scored on a six point ordinal scale, ranging from independent to dependent. Items can also be coded as participant refuses, not applicable, environmental limitations, not attempted due to medical condition or safety concerns, or unplanned discharge.
Manual Muscle Test | Baseline and Once weekly, through completion of study up to 4 weeks
  Manual Muscle Test is a procedure for evaluating the strength of 16 individual muscles relative to gravity and manual resistance. Instructions are provided to the participant before testing each muscle. A muscle is isolated, and gradual external force is applied at a right angle to the muscle's long axis. Each muscle is scored on a graded scale of "weak" to "strong" based on the participant's ability to resist the external force. The test is first completed for muscles on the unimpaired side to determine normal strength before being repeated on the impaired side. Weaker participants may be tested while lying prone (gravity eliminated).
Modified Ashworth Scale | Baseline and Once weekly, through completion of study up to 4 weeks
  The Modified Ashworth Scale is a 6-point ordinal scale used to grade the amount of hypertonicity in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
Step count | Each session, through completion of study up to 4 weeks
  The number of steps taken during each session will be measured using ActiGraph GT9X Link activity monitors. These devices are small accelerometers that can be worn on a belt and/or on the ankle to record steps and Kcals during an activity. The therapist leading the intervention session will apply the ActiGraph at the beginning of each intervention session and remove it upon completion.
Age-predicted maximum heart rate zone | Each session, through completion of study up to 4 weeks
  The target range of 70-85% of age-predicted maximum heart rate will be calculated for each participant utilizing HRmax = 208 - [0.7 × age] as developed by Tanka et al in 2001. It is recommended that clinicians should apply moderate to high-intensity walking training to improve walking speed and endurance individuals poststroke. The researchers will record the amount of time participants spend in their pre-calculated target zone during each gait training session utilizing the Polar OH1 Optical Heart Rate Sensor.
Borg Rating of Perceived Exertion | Baseline and Once weekly, through completion of study up to 4 weeks
  The Borg Rating of Perceived Exertion is a tool to measure the subjective report of effort, exertion, and fatigue during physical work. It consists of a 15-point scale from 6-20, in which 6=no exertion and 20=absolute maximum exertion. It is presented to the participant in written format with descriptors to standardize the report of perceived exertion across tasks.
Functional Gait Assessment (FGA) | Baseline and Once weekly, through completion of study up to 4 weeks
  The FGA is a 10-item test, scored on a four point ordinal scale. A higher score indicates decreased fall risk. It measures dynamic balance and postural stability during walking tasks (such as fast walking, backward walking, stepping over an obstacle) in the clinical setting. Patients are allowed to use an assistive device for certain items.
Passive Range of Motion | Baseline and Once weekly, through completion of study up to 4 weeks
  The purpose of this test is to evaluate a participant's passive range of motion in the joints of the hips, knees, and ankles. A larger range of motion indicates a better outcome.
Change in stride variability | Baseline and Once weekly, through completion of study up to 4 weeks
  Stride variability is the ratio between the standard-deviation and mean of stride time, expressed as percentage. Decreased variability indicates a better outcome.
Change in cadence | Baseline and Once weekly, through completion of study up to 4 weeks
  Cadence is the total number of steps taken within a given time period; often expressed per minute. Typically a higher number of steps is a better outcome.
Change in step length | Baseline and Once weekly, through completion of study up to 4 weeks
  Step length is the distance between the point of initial contact of one foot and the point of initial contact of the opposite foot. Typically a longer step length is a better outcome, ideally with equal measurements between left and right limbs.
Change in stride length | Baseline and Once weekly, through completion of study up to 4 weeks
  Between successive points of initial contact of the same foot. Right and left stride lengths are normally equal. Typically a longer stride length is a better outcome, ideally with equal measurements between left and right limbs.
Change in stance time | Baseline and Once weekly, through completion of study up to 4 weeks
  Stance time is the amount of time that passes during the stance phase of one extremity in a gait cycle. It includes single support and double support. Equal stance time between limbs is a better outcome.
Change in bilateral joint torque | Baseline and Once weekly, through completion of study up to 4 weeks
  Joint torque is the sum of passive and active torques of the human limb. Passive torques are produced by tension developed as muscle tissue, tendons, and ligaments are stretched. Active torque is the torque produced by the muscles. Typically lower joint torque during movement is a better outcome. This will be measured in the ankle, knee, and hip bilaterally

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No